CLINICAL TRIAL: NCT04374669
Title: The Influence of Sarcopenia on Outcomes of Neuroplasty in Patients With Lumbar Spinal Stenosis: a Prospective Observational Study
Brief Title: Sarcopenia and Outcomes of Neuroplasty in Lumbar Spinal Stenosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Doo-Hwan Kim, Assistant Professor, Asan Medical Center
Other Study IDs: S2020-0855-0001
Record Dates: First submitted 2020-04-24; First posted 2020-05-05 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Lumbar Spinal Stenosis; Neurogenic Claudication; Sarcopenia
Keywords: Sarcopenia; Frailty; Lumbar spinal stenosis; Neurogenic claudication; Neuroplasty
MeSH Terms: conditions — Spinal Stenosis; Sarcopenia; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with lumbar spinal stenosis: Patients with lumbar spinal stenosis will be scheduled for neuroplasty.
  Interventions: Procedure: Neuroplasty with Racz catheter

INTERVENTIONS:
Procedure: Neuroplasty with Racz catheter — The patient is placed in the prone position with a pillow placed under the abdomen to correct the lumbar lordosis. After sterile preparation and draping, the epidural space via the sacral hiatus using a 16 gauge needle is accessed. Then, the Racz catheter is advanced to the site of adhesions under the fluoroscopic guidance. The target site is determined by the location of pathology on lumbar MRI, preprocedural epidurography, and clinical symptoms before the adhesiolysis. Adhesiolysis is performed through the high-volume administration of medications, which consist of a combination of a steroid, local anesthetics, hyaluronidase, and 5% hypertonic saline. As needed, the catheter remains in the epidural space for two days, with the additional injection on each of the days.

SUMMARY:
The aim of the present study is to find out the influence of sarcopenia on outcomes of neuroplasty in patients with lumbar spinal stenosis.

DETAILED DESCRIPTION:
Frailty is an aging-related syndrome of physiological decline and correlated with sarcopenia. Furthermore, lumbar spinal stenosis is a common disease in the old population and a neuroplasty is widely used to treat these patients. We postulate that the sarcopenia may be associated with the outcome of neuroplasty in patients with lumbar spinal stenosis, and there is no study about this topic as far as we know.

To evaluate this association, we will use the criteria for sarcopenia which is made by Asian Working Group for Sarcopenia in 2019 in this study. We will compare the outcome of neuroplasty in patients with sarcopenia and without sarcopenia using several tools such as numeric rating scale (NRS), Oswestry Disability Index (ODI), and global perceived effect (GPE) score up to 6 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Presence of lumbar spinal stenosis on MRI
* 65 ≤ age <79
* Neurogenic claudication due to spinal stenosis
* Chronic pain above than 3 months despite conservative therapies
* Scheduled for neuroplasty with Racz catheter

Exclusion Criteria:

* Allergy to local anesthetics, contrast dye, or steroid
* Use of anticoagulants or antiplatelet medication
* Coagulopathy or Infection at the insertion site
* Neurological or psychiatric disorders
* Hemodynamic instability due to other underlying disorders
* Prior spine instrumentation
* Vascular claudication
* Refusal to participate in the study

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with lumbar spinal stenosis who is scheduled for neuroplasty in Asan medical center in Korea
Sampling Method: Non-Probability Sample
Enrollment: 79 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in numeric rating scale (NRS) at 3 months after the procedure | Before the procedure and 3 months after the procedure
  Numeric rating scale (0-10) 0=no pain, 10=worst pain imaginable
  We are going to compare the change of NRS at 3 months after the procedure to the baseline value.
Change in Oswestry disability index (ODI) at 3 months after the procedure | Before the procedure and 3 months after the procedure
  Oswestry disability index (10-60) 10: least score as possible, 60: most score as possible
  We are going to compare the change of ODI at 3 months after the procedure to the baseline value.
Global percieved effect (GPE) score at 3 months after the procedure | 3 months after the procedure
  Global percieved effect score by Likert scale (1-7)
  1: Never satisfied with the procedure, 7: Very satisfied with the procedure
Change in Medication Quantification scale (MQS) at 3 months after the procedure | Before the procedure and 3 months after the procedure
  Medication quantification scale is a tool to quantify medication regimen use in chronic pain populations. We are going to use Medication Quantification scale ver 3.
  The score starts at 0, and there is no specific maximum limit.
  We are going to compare the change of MQS at 3 months after the procedure to the baseline value.
The percentage of successful responders at 3 months after the procedure | 3 months after the procedure
  We are going to assess 4 variables above and then decide who is a successful responder or not at 3 months after the procedure.
  We defined the successful responders as follows;
  1. ≥ 50% or 4-point reduction from baseline leg Numeric rating scale and no increase from baseline Oswestry disability index and medication quantification scale and 4 points on the global perceived scale,
  2. ≥ 30% or 2 points reduction from baseline numeric rating scale with any one of the following criteria: simultaneous ≥ 30% (or 10-point) reduction in Oswestry disability index from baseline, or ≥ 5 points on global perceived effects scale, or no increase from the baseline medication quantification scale.
  NRS, ODI, and MQS will be evaluated before the procedure and become baseline values.
  NRS, ODI, and MQS will be re-evaluated, and GPE score will be newly evaluated 3 months after the procedure.

SECONDARY OUTCOMES:
Change in NRS at 1 and 6 months after the procedure | Before the procedure, and 1 and 6 months after the procedure
  We are going to compare the change of NRS at 1 and 6 months after the procedure to the baseline value.
Change in ODI at 1 and 6 months after the procedure | Before the procedure, and 1 and 6 months after the procedure
  We are going to compare the change of ODI at 1 and 6 months after the procedure to the baseline value.
GPE score at 1 and 6 months after the procedure | 1 and 6 months after the procedure
  We are going to check GPE score at 1 and 6 months after the procedure.
Change in MQS at 1 and 6 months after the procedure | Before the procedure, and 1 and 6 months after the procedure
  We are going to compare the change of MQS at 1 and 6 months after the procedure to the baseline value.
The percentage of successful responders at 1 and 6 months after the procedure | 1 and 6 months after the procedure
  We are going to evaluate successful responders at 1 and 6 months after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Doo-Hwan Kim, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bentov I, Kaplan SJ, Pham TN, Reed MJ. Frailty assessment: from clinical to radiological tools. Br J Anaesth. 2019 Jul;123(1):37-50. doi: 10.1016/j.bja.2019.03.034. Epub 2019 May 3. PMID 31056240
- [Background] Racz G, Candido K, Helm S. Neuroplasty Is a Safe, Effective Procedure. Anesth Analg. 2018 Jan;126(1):363. doi: 10.1213/ANE.0000000000002546. No abstract available. PMID 29135599
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Yamada Y, Nishizawa M, Uchiyama T, Kasahara Y, Shindo M, Miyachi M, Tanaka S. Developing and Validating an Age-Independent Equation Using Multi-Frequency Bioelectrical Impedance Analysis for Estimation of Appendicular Skeletal Muscle Mass and Establishing a Cutoff for Sarcopenia. Int J Environ Res Public Health. 2017 Jul 19;14(7):809. doi: 10.3390/ijerph14070809. PMID 28753945
- [Background] Choi SS, Lee JH, Kim D, Kim HK, Lee S, Song KJ, Park JK, Shim JH. Effectiveness and Factors Associated with Epidural Decompression and Adhesiolysis Using a Balloon-Inflatable Catheter in Chronic Lumbar Spinal Stenosis: 1-Year Follow-Up. Pain Med. 2016 Mar;17(3):476-487. doi: 10.1093/pm/pnv018. Epub 2015 Dec 7. PMID 26814254